CLINICAL TRIAL: NCT04685070
Title: Neoadjuvant HS-10296 (Almonertinib) Therapy for Potential Resectable Stage III EGFR Mutation-Positive Non-small Cell Lung Cancer: A Single-Arm, Open-Label, Phase II Clinical Trial
Brief Title: Neoadjuvant HS-10296 (Almonertinib) Therapy for Potential Resectable Stage III EGFR Mutation-Positive Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director of thoracic department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-007
Record Dates: First submitted 2020-12-05; First posted 2020-12-28 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Non-small Cell Lung Cancer Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10296 (Almonertinib) (Experimental)
  Interventions: Drug: HS-10296 (Almonertinib)

INTERVENTIONS:
Drug: HS-10296 (Almonertinib) — Neoadjuvant treatment stage: HS-10296 110mg, qd, po, 4 weeks per cycle, 2-4 cycles in total; Surgical treatment stage: CR + PR patients and SD + PD patients who could still undergo surgery will receive radical surgery; Adjuvant treatment stage: CR, PR and SD patients who have been treated surgically: HS-10296 110mg, qd, po, up to 48 weeks (including neoadjuvant stage). PD patients: transferred into medical oncology or/and radiation oncology and receive comprehensive therapy.

SUMMARY:
This is a phase II, single-arm, open-label study to evaluate the efficacy and safety of the third generation tyrosine kinase inhibitors (TKIs) Almonertinib (HS-10296) as neoadjuvant and adjuvant therapy for potential resectable stage III EGFR mutation-positive Non-small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC patient with EGFR sensitive mutation as confirmed by needle biopsy;
* At stage III (TNM Staging, Version 8) as identified by chest CT, PET-CT or/and EBUS;
* No systemic metastasis (confirmed by head MRI, whole body bone scan, PET-CT, liver and adrenal CT, etc.);
* With the feasibility to receive radical surgery ;
* Good lung function that could tolerate surgical treatment;
* Aged 18-75 years;
* At least one measurable tumor foci (the longest diameter measured by CT shall be > 10 mm);
* Other major organs shall function well (liver, kidney, blood system, etc.):
* ECOG PS score shall be 0-1;
* The child-bearing female must undergo pregnancy test within 7 days before starting the treatment and the result shall be negative. Reliable contraceptive measures, such as intrauterine device, contraceptive pill and condom, shall be adopted during the trial and within 30 days after completion of the trial. The child-bearing male shall use condom for contraception during the trial and within 30 days after completion of the trial;
* The patient shall sign the Informed Consent Form.

Exclusion Criteria:

* The patient has undergone any systemic anti-cancer treatment for NSCLC, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment, etc.;
* The patient suffered from other cancers besides NSCLC (except cervical carcinoma in situ, cured basal cell carcinoma and bladder epithelial tumor [including Ta and Tis]) within 5 years before the trial;
* The patient suffers from any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina pectoris, angina pectoris that starts to attack within the last 3 months, congestive heart failure [≥ Grade II specified by New York Heart Association (NYHA)], cardiac infarction (6 months before enrollment), severe arrhythmia and liver, kidney or metabolic diseases that requires drug treatment;
* The patient is a carrier of active hepatitis B, hepatitis C or HIV;
* The patient suffers from severe or new-onset gastrointestinal diseases with diarrhea as the main symptom;
* The patient has had or is currently suffering from cardiovascular malformation;
* The patient has had or is currently suffering from interstitial lung disease;
* The patient had undergone other major systemic operations or suffered from severe trauma within 3 months before the trial;
* The patient is allergic to afatinib or its any excipients;
* The patient suffers from nervous system diseases or mental diseases and cannot keep compliance with the trial;
* The patient has any malabsorption condition;
* The female patient is in pregnancy or lactation period;
* There are any conditions under which the investigator considers the patient is not suitable to be enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 4 months
  ORR is defined as the proportion of patients who have completed the neoadjuvant treatment before operation and have achieved CR or PR as confirmed by CT evaluation in all patients.

SECONDARY OUTCOMES:
Major pathologic response (MPR) | up to 5 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery.
Event free survival (EFS) | up to 60 months
  It refers to the time from randomization to disease progression, cessation of treatment for any reason, or death
Overall survival (OS) | up to 60 months
  It is defined as the time from random enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
R0 resection rate | up to 6 months
  complete removal of the tumor, with a negative microscopic margin indicating no residual tumor
Treatment-related adverse events | up to 13 months
  It refers to the number of adverse events related to HS-10296 as evaluated according to CTCAE v4.0.
Pathological complete response rate (pCR) | up to 24 months
  It refers to the number of cases with no residual invasive cancer in the primary tumor and lymph node HE staining accounted for the proportion of all patients who completed the treatment.

OTHER OUTCOMES:
Potential biomarkers | up to 24 months
Tumor microenvironment dynamics | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided